CLINICAL TRIAL: NCT05563948
Title: Repeated Administration of Cannabis Varying in THC and CBD: Effects on Abuse Liability, Experimental Pain and Plasma Endocannabinoids
Brief Title: Repeated Administration of Cannabis Varying in THC and CBD
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: In response to quality assurance and compliance concerns, OHRP issued an FWA restriction on NYSPI research that included a pause of human research as of June 23, 2023.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Margaret Haney, Clinical professor in Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 8347
Record Dates: First submitted 2022-09-26; First posted 2022-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- High THC : High CBD (Experimental): Cannabis that is high in THC and high in CBD will be administered.
  Interventions: Drug: Cannabis
- High THC : Low CBD (Experimental): Cannabis that is high in THC and low in CBD will be administered.
  Interventions: Drug: Cannabis
- Low THC : High CBD (Experimental): Cannabis that is low in THC and high in CBD will be administered.
  Interventions: Drug: Cannabis
- Low THC : Low CBD (Placebo Comparator): Cannabis that is low in THC and low in CBD will be administered.
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — Vaporized cannabis will be administered 3x/day for 15 days.

SUMMARY:
The majority of the >3 million medical cannabis patients in the U.S. use cannabis products to manage pain but many questions remain. This project is designed to answer three questions that will fill important voids in the field's understanding of sustained cannabis use: 1) is abrupt cessation of cannabis associated with increased pain sensitivity; 2) does tolerance develop to the analgesic and abuse-related effects of repeatedly administered cannabis with varying ratios of THC and CBD, and is this tolerance reversible following a period of abstinence; 3) how does repeated cannabis use affect levels of endocannabinoids, and are these changes associated with changes in pain sensitivity and abuse liability? In this study, the investigators will enroll participants (N=100 healthy, cannabis-using men and non-pregnant women, ages 21-65) inpatient for 15 days. They will be randomized to one of four cannabis conditions (n=25/group). Following a day of standardization on which participants will receive their assigned cannabis condition (Day 1), cannabis will be administered repeatedly for 14 days (Day 2-15). The investigators will measure abuse-related effects ("Good Drug Effect"), endocannabinoid levels and two distinct types of experimental pain: The Cold Pressor Test and Quantitative Sensory Testing Thermal Temporal Summation. Given the widespread use of cannabis for pain, understanding the consequences of daily repeated administration of cannabis with THC:CBD ratios that are representative of most medical cannabis products on pain, abuse liability, and endocannabinoids is imperative.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 21-65 years old
2. For females: not pregnant or breast-feeding, and uses an acceptable form of birth control (e.g., condoms, IUD)
3. Uses cannabis on a near-daily basis
4. Not seeking treatment for cannabis use
5. Able to provide informed consent
6. Able to perform study procedures

Exclusion Criteria:

1. Meets DSM-V criteria for any Substance Use Disorder other than cannabis, nicotine or caffeine
2. Uses other illicit drugs ≥1 day/week in the prior 4 weeks
3. Medical history, physical, psychiatric examination, or significant illness at the clinical discretion of the study physician; for example, history of heart disease, diabetes, hypertension (BP > 140/90) or uncontrolled asthma

5. Use of any prescription or daily use of over-the-counter medications 6. Recurrent, ongoing pain 7. Insensitivity to the thermal stimuli of the Cold Pressor Test or Quantitative Sensory Testing 8. History of physical violence or paranoia during cannabis withdrawal

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2032-09-30 (Estimated); Study Completion 2034-09-30 (Estimated)

PRIMARY OUTCOMES:
Cold Pressor Test (Change over time from baseline) | 8x/day on Days 1, 2, 5, 8, 9, 12, 15.
  The Cold Pressor Test (CPT) is a validated and reliable pain-induction procedure that reflects A-delta nerve fiber activity within the autonomic nervous system and closely mimics clinical chronic pain. CPT has been shown to have excellent reliability and predictive validity for medication-induced analgesia, including cannabinoids. For this task, two temperature-controlled circulating water baths maintain warm (36.5-37.5ºC) and cold (3.5-4.5ºC) water. Participants immerse their hand into a warm bath for 3 min (to standardize baseline skin temperature), then the cold bath, indicating when they first experience pain and withdrawing when the pain gets uncomfortable. Study staff will record time (in seconds) until participants: 1) report discomfort (pain threshold), and 2) withdraw their hand from the cold water (pain tolerance).
Quantitative Sensory Testing-Thermal Temporal Summation (QST-TTS; change over time from baseline) | 8x/day on Days 1, 2, 5, 8, 9, 12, 15.
  (QST-TTS) uses repetitive fixed frequency and intensity heat stimulation to induce central sensitization of C-fibers in the spinal cord and is regarded as an experimental correlate of the 'wind-up' phenomenon in the dorsal horn. As dorsal horn CB-1 activity has been linked to suppression of 'wind-up' and central sensitization (the mechanism purportedly underlying cannabis' efficacy for neuropathic pain), cannabis use may decrease QST-TTS response, mirroring analgesia on the CPT during active cannabis administration vs. placebo. For this task, a Medoc TSA-II NeuroSensory Analyzer with a 30 x 30 mm Peltier thermode applies tonic noxious heat stimulation to the thenar eminence of the palm: the baseline temperature is 32.0°C, increases at a rate of 1°C/s up to 46.5°C, and remains constant for 120 sec. Total duration.

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided